CLINICAL TRIAL: NCT01880580
Title: Cone Beam CT for Breast Imaging: A Pilot Study
Brief Title: Cone Beam CT for Breast Imaging
Status: Completed | Type: Observational
Sponsor: Koning Corporation (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: URMC-001
Record Dates: First submitted 2013-06-15; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Breast Imaging; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal Group: In Group I, up to 100 women, at least 40 years of age, who have had a routine standard mammogram read as BI-RADS® 0, 1, 2, or 3 will also undergo 3D breast imaging using a cone beam CT scanner specifically designed to image the breast. Of these 100, we hope to enroll at least 30 subjects with mammograms read as BI-RADS® 0 and at least 30 read as BI-RADS® 3. The BI-RADS® 0 category refers to patients for whom additional imaging is required after a screening mammogram provided incomplete diagnostic information.
- Diagnostic Group: The goals of Group II will be to compare the CBCT study with standard imaging for the diagnosis of breast disease in palpable or non-palpable breast lesions (having a BI-RADS® score of 4 or 5). Forty (40) women, who have had abnormalities detected by physical exam or an imaging modality and are also scheduled for breast biopsy of the index lesion, will also undergo a CBCT of the breast(s), prior to biopsy.

SUMMARY:
The objective of this pilot study is to investigate Cone Beam Computed Tomography Imaging (CBCT), with the primary goal, the accumulation of a body of evidence to provide preliminary data for a future extensive clinical trials.

ELIGIBILITY:
Normal Group:

Inclusion Criteria:

* Are at least 40 years of age of any ethnicity
* Had a routine mammogram, read as BI-RADS® 0, 1, 2 or 3
* Will undergo study imaging no later than six months from date of routine mammogram.
* Is able to undergo informed consent.

Exclusion Criteria:

* Pregnancy
* Lactation
* Patients with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Patients who are unable to tolerate study constraints.
* Patients who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkin's disease
* Patients who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Patients who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis

Diagnostic Group:

Inclusion Criteria:

* Women who are at least 40 years of age of any ethnicity
* Have a palpable abnormality detected by Breast Self Exam (BSE), or Clinical Breast Exam (CBE) or have a non-palpable abnormality detected by an imaging modality
* After diagnostic work-up are categorized as BI-RADS® 4 or 5.
* Are scheduled for biopsy either by large gauge needle biopsy or excisional biopsy.
* Will undergo study imaging prior to biopsy and within four weeks of diagnostic work-up.

Exclusion Criteria:

* Pregnancy
* Lactation
* Patients who have already undergone biopsy for the index lesion
* Patients who are unable or unwilling to undergo biopsy for the lesion of concern
* Patients with physical limitations that may prohibit the patient from resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Patients who are unable to tolerate study constraints.
* Patients who have received radiation treatments to the thorax or breast area for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkin's disease
* Patients who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Patients who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In Group I, up to 100 women, at least 40 years of age, who have had a routine standard mammogram read as BI-RADS® 0, 1, 2, or 3 will also undergo 3D breast imaging using a cone beam CT scanner specifically designed to image the breast.
  Group II includes forty (40) women, who have had abnormalities detected by physical exam or an imaging modality and are also scheduled for breast biopsy of the index lesion, will also undergo a CBCT of the breast(s), prior to biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2006-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Image Quality of Cone Beam Breast CT | 6 years
  This study was to evaluate the radiation dose, breast coverage, and image quality of cone-beam breast CT compared with a conventional mammographic examination.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Highland Breast Imaging Center, Rochester, New York, United States

REFERENCES:
- [Result] O'Connell A, Conover DL, Zhang Y, Seifert P, Logan-Young W, Lin CF, Sahler L, Ning R. Cone-beam CT for breast imaging: Radiation dose, breast coverage, and image quality. AJR Am J Roentgenol. 2010 Aug;195(2):496-509. doi: 10.2214/AJR.08.1017. PMID 20651210
- [Result] O'Connell AM, Kawakyu-O'Connor D. Dedicated Cone-beam Breast Computed Tomography and Diagnostic Mammography: Comparison of Radiation Dose, Patient Comfort, And Qualitative Review of Imaging Findings in BI-RADS 4 and 5 Lesions. J Clin Imaging Sci. 2012;2:7. doi: 10.4103/2156-7514.93274. Epub 2012 Feb 25. PMID 22439131